CLINICAL TRIAL: NCT07344064
Title: The Effects of Adjunctive Therapy With Vaginal Tablets Lactobacillus Acidophilus and a Low Dose Estriol (Gynoflor®) to Prolong Pregnancy Time in Preterm Labor, A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 015/2568
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Threaten Preterm; Prethrem Labour; Bacterial Vaginitis
Keywords: Lactobacillus; Gynoflor; Threaten preterm; Bacterial vaginitis; Probiotic
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- gynoflor group (Experimental)
  Interventions: Drug: Gynoflor
- control group (No Intervention)

INTERVENTIONS:
Drug: Gynoflor — Participants in this group will receive Gynoflor vaginal tablets (containing Lactobacillus acidophilus and estriol) administered once daily for 7 consecutive days. This intervention aims to evaluate whether restoring vaginal flora with Gynoflor can prolong pregnancy time compared to no intervention.
  Arms: gynoflor group

SUMMARY:
The study aim to study The Adjunctive therapy with vaginal tablets containing Lactobacillus acidophilus KS400 and low-dose Estriol (Gynoflor®) in addition to standard tocolytic treatment administered once daily for 6 days starting the same day as tocolytic therapy, in pregnant women diagnosed with preterm labor at gestational age 24-33 weeks .Primary Outcome is the rate of pregnancy prolongation beyond 7 days after initiation of tocolytic therapy.

DETAILED DESCRIPTION:
Participants in the intervention group are pregnant women diagnosed with preterm labor between 24 and 33 weeks of gestation. They receive:

* Gynoflor® vaginal tablets (containing Lactobacillus acidophilus KS400 and 0.03 mg estriol)
* Dosage: 1 tablet inserted vaginally at bedtime for 6 consecutive days
* Start time: On the same day as starting standard tocolytic therapy (such as nifedipine, terbutaline, or magnesium sulfate)
* Purpose: To restore healthy vaginal flora, reduce risk of ascending infection, and potentially prolong pregnancy duration

The control group receives only standard tocolytic therapy, without Gynoflor®.

Outcomes (Detailed Description):

Primary Outcome:

* Rate of pregnancy prolongation beyond 7 days from the initiation of tocolytic therapy

Secondary Outcomes:

1. Gestational age at delivery ≥34 weeks
2. Length of hospital stay (in days)
3. Use of second-line tocolytic agents (e.g., switching due to inefficacy or side effects)
4. Readmission within 14 days after discharge
5. Incidence of side effects from Gynoflor® (especially local symptoms like vaginal burning or irritation)

ELIGIBILITY:
Inclusion Criteria

- Pregnant women diagnosed with preterm labor or threatened preterm labor, with a gestational age between 24 and 33 weeks, who are receiving tocolytic therapy.

Exclusion Criteria

* Age under 18 years or 35 years and older
* Incomplete course of Gynoflor® (less than 6 days of use)
* Presence of contraindications to tocolysis
* Preterm premature rupture of membranes (PPROM)
* Unable to be contacted for follow-up
* History of allergy to probiotics or Gynoflor®
* Multiple gestation
* History of short cervix diagnosed between 16-24 weeks of gestation
* History of previous preterm labor (PTL)
* Pregnancy achieved via assisted reproductive technology (ART)
* Presence of fetal anomaly
* History of antepartum hemorrhage
* Substance abuse, including cigarette smoking, alcohol, cocaine, or heroin use
* Other causes of preterm labor such as uterine overdistension (e.g., polyhydramnios, multifetal gestation), uterine abnormalities (e.g., myoma uteri), or systemic infections, except vaginitis

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
proportion of women remaining pregnant more than 7 days after initiation of tocolytic | within 7 days from the start of tocolytic

IPD SHARING:
Plan to Share IPD: Yes